CLINICAL TRIAL: NCT04317183
Title: The Effect of Topical Chamomile in the Prevention of Chemotherapy-induced Oral Mucositis (a Randomized Controlled Clinical Trial)
Brief Title: Topical Chamomile in Preventing Chemotherapy-induced Oral Mucositis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00010556-IORG 0008839
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Oral Mucositis Due to Chemotherapy
Keywords: oral mucositis, chemotherapy, chamomile.
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chamomile topical gel (Experimental): Topical oral chamomile gel three times daily for three weeks.
  Topical oral chamomile gel is prepared with the aid of Pharmacognosy and pharmaceutics departments, faculty of pharmacy, Alexandria University and mucoadhesive hydrogels (Carbopol® 970).
  Interventions: Drug: chamomile topical oral gel
- conventional therapy (Active Comparator): Conventional therapy (symptomatic treatment) which included:
  Miconaz oral gel BBC oral spray Oracure gel
  Dose: Three times a day for three weeks
  Interventions: Drug: Miconazole Topical Gel; Drug: BBC oral spray; Drug: Oracure gel
- combination therapy (Experimental): Topical oral chamomile gel three times daily for three weeks in combination with the symptomatic treatment
  Symptomatic treatment which included:
  Miconaz oral gel BBC oral spray Oracure gel
  Symptomatic treatment dose: Three times a day for three weeks
  Interventions: Drug: chamomile topical oral gel; Drug: Miconazole Topical Gel; Drug: BBC oral spray; Drug: Oracure gel

INTERVENTIONS:
Drug: chamomile topical oral gel — Chemical constituents of chamomile, such as bisabolol, chamazulene, and the flavonoids apigenin and luteolin, possess anti-inflammatory properties.
  Arms: Chamomile topical gel; combination therapy
Drug: Miconazole Topical Gel — topical anti fungal agent
  Arms: combination therapy; conventional therapy
Drug: BBC oral spray — Topical anesthetics and anti-inflammatory agent
  Arms: combination therapy; conventional therapy
Drug: Oracure gel — Topical analgesic gel
  Arms: combination therapy; conventional therapy

SUMMARY:
the main aim of this study is to clinically assess the effectiveness of topical chamomile oral gel in the prevention of chemotherapy-induced oral mucositis.

DETAILED DESCRIPTION:
The study was designed as a randomized, controlled, clinical trial. patients who were undergoing to receive chemotherapy were divided into three groups: Group I: was given conventional treatment. Group II: was given topical oral gel of chamomile. Group III: was given topical oral gel of chamomile in combination with the conventional treatment.

All patients have clinically evaluated at the start of the chemotherapy and three weeks later for pain and oral mucositis severity.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are going to receive 5-Fluoroucil (5-FU) based chemotherapy regime.

Males and females with an age of not less than 20 years and not exceeding 70 years.

Exclusion Criteria:

* 1. Patients suffering from any uncontrolled systemic diseases that affect integrity of the epithelium (such as diabetes, cardiovascular, liver disorder and renal dysfunction) 2. Pregnant and lactating women 3. Patients with findings of any physical or mental abnormality which would interfere with or be affected by the study procedure

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Changes in severity of oral mucositis at different time points along the study | Up to 3 weeks
  Oral mucositis will be evaluated by the World Health Organization (WHO) scale which record the extent and severity of oral mucositis at the third week after the first chemotherapy session.

SECONDARY OUTCOMES:
Pain and discomfort severity at different time points along the study: Numeric Rating Scale | Up to 3 weeks
  Discomfort and pain severity were reported by each patient using Numeric Rating Scale (NRS) at the first , second and third week after the chemotherapy session.

CONTACTS AND LOCATIONS:
Overall Officials: Ehsan El-Negomy, PhD, Study Director — Alexandria University; Maha Talaab, PhD, Study Director — Alexandria University; Reham Ibrahim, Phd, Study Director — Alexandria University; Rasha El-Saka, Study Director — Alexandria University
Locations (1):
- Outpatient clinic of Department of Clinical Oncology, Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Presibella MM, Villas-Bôas LDB, Belletti KMdS, Santos CAdM, Weffort-Santos AM. Comparison of chemical constituents of Chamomilla recutita (L.) Rauschert essential oil and its anti-chemotactic activity. Brazilian archives of biology and technology. 2006;49(5):717-24.
- [Background] Ferreira E, Vasques C, Jesus C, Reis P. Topical effects of Chamomilla recutita in skin damage: a literature review. 2015.
- [Background] Tadbir AA, Pourshahidi S, Ebrahimi H, Hajipour Z, Memarzade MR, Shirazian SJJoHM. The effect of Matricaria chamomilla (chamomile) extract in Orabase on minor aphthous stomatitis, a randomized clinical trial. 2015;5(2):71-6.
- [Background] Fidler P, Loprinzi CL, O'Fallon JR, Leitch JM, Lee JK, Hayes DL, Novotny P, Clemens-Schutjer D, Bartel J, Michalak JC. Prospective evaluation of a chamomile mouthwash for prevention of 5-FU-induced oral mucositis. Cancer. 1996 Feb 1;77(3):522-5. doi: 10.1002/(SICI)1097-0142(19960201)77:33.0.CO;2-6. PMID 8630960
- [Background] Braga FT, Santos AC, Bueno PC, Silveira RC, Santos CB, Bastos JK, Carvalho EC. Use of Chamomilla recutita in the Prevention and Treatment of Oral Mucositis in Patients Undergoing Hematopoietic Stem Cell Transplantation: A Randomized, Controlled, Phase II Clinical Trial. Cancer Nurs. 2015 Jul-Aug;38(4):322-9. doi: 10.1097/NCC.0000000000000194. PMID 25232958
- [Background] Baydar M, Dikilitas M, Sevinc A, Aydogdu I. Prevention of oral mucositis due to 5-fluorouracil treatment with oral cryotherapy. J Natl Med Assoc. 2005 Aug;97(8):1161-4. PMID 16173332
- [Background] Sonis ST, Elting LS, Keefe D, Peterson DE, Schubert M, Hauer-Jensen M, Bekele BN, Raber-Durlacher J, Donnelly JP, Rubenstein EB; Mucositis Study Section of the Multinational Association for Supportive Care in Cancer; International Society for Oral Oncology. Perspectives on cancer therapy-induced mucosal injury: pathogenesis, measurement, epidemiology, and consequences for patients. Cancer. 2004 May 1;100(9 Suppl):1995-2025. doi: 10.1002/cncr.20162. PMID 15108222
- [Background] Rubenstein EB, Peterson DE, Schubert M, Keefe D, McGuire D, Epstein J, Elting LS, Fox PC, Cooksley C, Sonis ST; Mucositis Study Section of the Multinational Association for Supportive Care in Cancer; International Society for Oral Oncology. Clinical practice guidelines for the prevention and treatment of cancer therapy-induced oral and gastrointestinal mucositis. Cancer. 2004 May 1;100(9 Suppl):2026-46. doi: 10.1002/cncr.20163. PMID 15108223